CLINICAL TRIAL: NCT05055037
Title: Exploring the Feasibility of Neurofeedback for Trauma-affected Refugees - a Qualitative Study
Brief Title: Neurofeedback as a Treatment for Trauma-affected Refugees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Lundbeck Foundation (Other); Jascha Fonden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NF
Record Dates: First submitted 2021-07-26; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-07

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Neurofeedback; Refugee; Trauma; Qualitative study
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neurofeedback — In neurofeedback (NF), the brainwave activity is measured by an electro-encephalography and fed back to the person as an auditory or visual signal, rewarding the person each time progress is made toward normalizing dysregulated neural activity. The learning mechanism is at its base considered to be operant conditioning, where the behavior of the participant-in this case, neurological activity-is gradually changed through repeated reinforcement. In neurofeedback, this simple learning mechanism is accelerated by continuous and instant feedback, with rewards occurring as often as every second. The NF intervention included 12 NF training sessions, one session per week, off approximately 12-20 min. The protocol was a replicate of the setup of recent NF studies investigating NF as a treatment for chronic PTSD. The feedback was based on a single channel recording, rewarding brainwave frequencies associated with a calm and relaxed state and inhibiting drowsiness and hyperarousal.

SUMMARY:
Neurofeedback (NF) is a form of treatment that can assist individuals in learning to control their brain wave activity. NF-studies have shown promising results in reducing PSTD-symptoms among military veterans, but there are no published peer-reviewed studies with refugees. However, preliminary studies from Malmö and Sydney indicate that refugees could benefit from NF. Therefore, at the Competence Centre for Transcultural Psychiatry (CTP) a longitudinal feasibility study, testing NF for trauma-affected was started. The study contains both a quantitative and a qualitative substudy. In in the quantitative substudy, where a total of 32 participants have been included, the aim was to evaluate the feasibility of NF with trauma affected refugees using a quantitative perspective. The NF intervention offered was 12 training sessions of 12-20 minutes NF, and the outcome measures were self-administered questionnaires and semi-structured interviews collected before and after the intervention. In a subsample of eight participants of those included in the quantitative substudy, qualitative in-depth interviews were carried out. The participants were offered two interviews; one before the first NF training and one during the treatment course. The aim of the qualitative substudy was to evaluate the feasibility of NF with trauma-affected refugees by examining the participants' thoughts and expectations prior to participating in NF treatment as well as their experience with the treatment after a few sessions.

ELIGIBILITY:
Inclusion Criteria:

* Refugee or a person who had been family reunified with a refugee
* Diagnosed with PTSD (ICD-10 diagnosis F43.1) and experienced a psychological trauma in another country than Denmark.
* Informed consent.

Exclusion Criteria:

* Current abuse of drug or alcohol (F1x.24-F1x.26)
* Diagnosed with a severe psychotic disorder (F2x) or a manic disorder (F30.1-F31.9).
* No informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Harvard Trauma Questionnaire (HTQ) | Baseline and after 12 weeks
  Change in PTSD symptoms measured by the first 16 items in the Harvard Trauma Questionnaire

SECONDARY OUTCOMES:
Hopkins Symptom Checklist-25 (HSCL-25) | Baseline and after 12 weeks
  Change in depressive and anxiety symptoms
Sheehan Disability Scale (SDS) | Baseline and after 12 weeks
  Changes in functioning
WHO-Five Well-being Index (WHO-5) | Baseline and after 12 weeks
  Change in quality of life
Hamilton interview-based rating scales for depression (Ham-D) and anxiety (Ham-A) | Baseline and after 12 weeks
  Change in depressive and anxiety symptoms
Satisfaction and Accept-ability Questionnaire (SAQ) | After 12 weeks
  Evaluation of the the patients' satisfaction and potential discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Z Hannemose, MD, Principal Investigator — Competence Centre for Transcultural Psychiatry
Locations (1):
- Competence Centre for Transcultural Psychiatry, Ballerup Municipality, Denmark

REFERENCES:
- [Derived] Hannemose SZ, Laugesen Attardo H, Vindbjerg E, Carlsson J. Exploring expectations of neurofeedback treatment among trauma-affected refugees. Nord J Psychiatry. 2024 Jan;78(1):46-53. doi: 10.1080/08039488.2023.2261905. Epub 2024 Jan 8. PMID 37755151
- See also: Description Link to web page of the Competence Centre for Transcultural Psychiatry (mostly in Danish) — https://www.psykiatri-regionh.dk/centre-og-social-tilbud/kompetencecentre/transkulturel-psykiatri/Sider/default.aspx